CLINICAL TRIAL: NCT01683734
Title: Nephrotoxicity Following 2-Stage Exchange With Associated Antibiotic Laden Spacer in Patients With Infected Total Hip/Knee Arthroplasty
Brief Title: Assessing Renal Function in Patients With an Antibiotic Laden Spacer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central DuPage Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Nephro11-021-1
Record Dates: First submitted 2012-08-28; First posted 2012-09-12 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Infected Total Hip or Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Function Observation

SUMMARY:
The purpose of this study is to monitor the renal function of patients who have an antibiotic laden spacer in place to treat an infected hip or knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing a hip or knee resection arthroplasty by the primary investigator
2. Ages 18+
3. Ability to adhere to follow up schedule

Exclusion Criteria:

1. Unable to give informed consent
2. Age <18
3. Previous history of infected Total Knee Arthroplasty or Total Hip Arthroplasty
4. History of renal failure or impaired renal function
5. Allergies to aminoglycosides or Vancomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with an infected hip or knee arthroplasty scheduled to undergo a 2-stage resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Development of acute renal insufficiency or acute renal failure measured by changes in laboratory values assessing renal function | subjects will be followed during the time the antibiotic spacer is in place which is approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sporer, MD, Principal Investigator — RUSH University Medical Center; Central DuPage Hospital
Locations (2):
- United States (2):
  - RUSH University Medical Center, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois